CLINICAL TRIAL: NCT05971147
Title: Time Course Change in Skeletal Muscle and Blood Phospholipid Composition With Omega-3 Fatty Acid Supplementation and Washout in Adult Women and Men
Brief Title: Time Course Change in Skeletal Muscle and Blood Phospholipid Composition With Omega-3 Fatty Acid Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Chris McGlory, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Chris McGlory, PhD, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6037330
Record Dates: First submitted 2023-07-18; First posted 2023-08-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-01

CONDITIONS: Skeletal Muscle Fatty Acid Metabolism
Keywords: Omega-3 fatty acids; Eicosapentaenoic acid; Docosahexaenoic acid; Fish oil; Skeletal muscle
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Single-arm 5g per day of omega-3 fatty acid intake (3750 mg EPA and 1250 mg DHA)
Masking Description: All participants will take part in the same intervention, which will be fully disclosed to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fish Oil Group (Experimental): All participants will be placed in this group
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil — Participants in this group will receive 5g fish oil with high EPA and DHA content per day

SUMMARY:
Increased omega-3 fatty acid composition of human skeletal muscle phospholipids is linked to improved skeletal muscle strength and growth in women and men. However, what is unknown is if biological sex influences skeletal muscle phospholipid composition in response to omega-3 fatty acid supplementation. Moreover, whilst time course changes in skeletal muscle phospholipid composition with omega-3 fatty acid intake have been established, no study has characterized a washout of omega-3 fatty acids from skeletal muscle phospholipids following cessation of omega-3 fatty acid intake. Thus, the aim of the present investigation is to establish a time course change and washout of omega-3 fatty acids from skeletal muscle phospholipids in response to omega-3 fatty acid intake. The investigators also aim to establish if this washout is impacted by biological sex.

DETAILED DESCRIPTION:
Previous work has shown that supplementing with omega-3 fatty acids leads to increased omega-3 fatty acid composition of skeletal muscle phospholipids. This increase in skeletal muscle omega-3 fatty acid phospholipid composition following omega-3 fatty acid intake is linked to potentiated rates of skeletal muscle protein synthesis in response to amino acid and insulin infusion in older and younger women and men. Supplementation with omega-3 fatty acids is also known to enhance skeletal muscle strength and size in older adults. The exact biological mechanisms responsible for the anabolic influence of omega-3 fatty acid are unknown. However, there is emerging data that acid (EPA) and docosahexaenoic acid (DHA) play an active role. Indeed, there is now a growing body of evidence in cells, preclinical models, and humans that these key omega-3 fatty acids are primarily responsible for the observed anabolic impact of omega-3 fatty acids supplement intake towards skeletal muscle.

Whilst there is a growing body of literature supporting the anabolic potential of EPA and DHA in skeletal muscle, few studies have examined how biological sex influences EPA and DHA incorporation into skeletal muscle. Indeed, it has been purported that women EPA to DHA more efficiently in blood erythrocytes compared to men. To the investigators knowledge, no study examined how biological sex impacts changes in skeletal muscle phospholipid profiles in response to EPA and DHA intake. Moreover, no study has established a time course washout of EPA and DHA from skeletal muscle phospholipids in response to the cessation of EPA and DHA intake. The lack of data regarding EPA and DHA washout from skeletal muscle in response to EPA and DHA intake limits the ability to execute within subject cross over trials, which is important given that within-subject cross over trials possess more statistical power than parallel arm trials. Thus, establishing a washout of EPA and DHA from skeletal muscle phospholipids in response to EPA and DHA intake would provide important information for the design of future trials in this field.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-30 years
* BMI between 18-29 kg/m2
* Free of musculoskeletal injuries
* Participants not currently pregnant
* Participants willing to maintain current use of contraceptives or post-menopausal supplementation if any for the duration of the study.
* Not allergic to fish
* COVID-19 vaccinated to comply with Queen's University's return to campus guidelines, unless exempt by reasons from the Ontario Human Rights Code
* Recreationally active

Exclusion Criteria:

* Any muscular, neurological, respiratory or metabolic disease including diabetes
* Any form of cancer currently or in the last 5 years
* Currently taking fish oil supplements
* Currently taking any form of steroid
* Consuming >2 oily fish meals per week
* Pregnant
* Any current illness
* Any current/past lower limb injury/surgery

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Changes in skeletal muscle EPA and DHA content | At 0, 6, 8, 16, 20, and 22 weeks.
  Skeletal muscle phospholipid composition will be assessed at all time points by means of gas chromatography

SECONDARY OUTCOMES:
Changes in the expression of mitochondrial related proteins | 0, 6, 8, 16, 20, and 22 weeks.
  Mitochondrial proteins involved in oxidative phosphorylation (e.g. ANT1) will be assessed by means of western blotting at all time points.
Changes in erythrocyte EPA and DHA content | 0, 6, 8, 16, 20, and 22 weeks.
  Erythrocyte phospholipid composition will be assessed at all time points by means of gas chromatography
Changes in the expression of translational factors related to skeletal muscle protein synthesis | 0, 6, 8, 16, 20, and 22 weeks.
  Translational factors involved in skeletal muscle protein synthesis (e.g. p70S6K1) will be assessed by means of western blotting at all time points.
Changes in circulating glucose concentrations | 0, 6, 8, 16, 20, and 22 weeks.
  Glucose concentrations will be assessed by ELISA at all time points.
Changes in circulating insulin concentrations | 0, 6, 8, 16, 20, and 22 weeks.
  Insulin concentrations will be assessed by ELISA at all time points.
Changes in circulating TNFa concentrations | 0, 6, 8, 16, 20, and 22 weeks.
  TNFa concentrations will be assessed by ELISA at all time points.
Changes in circulating CRP concentrations | 0, 6, 8, 16, 20, and 22 weeks.
  CRP concentrations will be assessed by ELISA at all time points.

CONTACTS AND LOCATIONS:
Overall Officials: Chris McGlory, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Health Studies, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be retained by the investigators, and shared under reasonable request.